CLINICAL TRIAL: NCT07360756
Title: Early Prediction of Post-Dural Puncture Headache Using Ultrasound-Measured Optic Nerve Sheath Diameter in Cesarean Section Patients: A Prospective Observational Study
Brief Title: Ultrasonographic ONSD as a Predictor of PDPH in Spinal Anesthesia for Cesarean Delivery
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Other Study IDs: RC. 1.12.2025
Record Dates: First submitted 2025-12-26; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Section Complications
Keywords: Post-Dural Puncture Headache; Optic Nerve Sheath Diameter
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort (Single Cohort): This study comprises a single, prospectively enrolled cohort of 150 adult female patients (ASA physical status II-III) scheduled for elective cesarean section under standardized spinal anesthesia. All participants receive the same planned intervention (spinal anesthesia for surgery) and undergo the same standardized measurement protocol for Optic Nerve Sheath Diameter (ONSD). Within this cohort, participants are naturally divided by outcome during follow-up into two groups for analytical purposes:
  PDPH-Positive Subgroup: Patients who develop Post-Dural Puncture Headache (PDPH) within 72 hours, as diagnosed using the International Classification of Headache Disorders (ICHD-3) criteria.
  PDPH-Negative Subgroup: Patients who do not develop PDPH within the follow-up period.
  Interventions: Procedure: Study Cohort (Single Cohort)

INTERVENTIONS:
Procedure: Study Cohort (Single Cohort) — This study comprises a single, prospectively enrolled cohort of 150 adult female patients (ASA physical status II-III) scheduled for elective cesarean section under standardized spinal anesthesia. All participants receive the same planned intervention (spinal anesthesia for surgery) and undergo the same standardized measurement protocol for Optic Nerve Sheath Diameter (ONSD). Within this cohort, participants are naturally divided by outcome during follow-up into two groups for analytical purposes:
  PDPH-Positive Subgroup: Patients who develop Post-Dural Puncture Headache (PDPH) within 72 hours, as diagnosed using the International Classification of Headache Disorders (ICHD-3) criteria.
  PDPH-Negative Subgroup: Patients who do not develop PDPH within the follow-up period.

SUMMARY:
The Optic Nerve Sheath Diameter (ONSD), measured non-invasively by bedside ultrasound, is a well-established surrogate for intracranial pressure (ICP), as the optic nerve sheath is continuous with the intracranial dura mater and its subarachnoid space is filled with cerebrospinal fluid (CSF). While ONSD is typically used to detect elevated ICP (with a cut-off often > 5.0-5.7 mm for ICP > 20 mmHg), studies investigating PDPH have paradoxically shown a reduction in ONSD post-spinal anesthesia, correlating with the state of intracranial hypotension.

Previous research has demonstrated that a lower ONSD or a significant decrease in ONSD values 24 hours post-puncture is associated with PDPH development. A study determined that an ONSD at 24 hours of less than 0.40 cm was the best predictor for PDPH. Our study aims to specifically investigate the utility of the immediate change in ONSD to offer a bedside, real-time assessment of risk.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients, aged 18-45 years
* ASA(American Society of Anesthesiologists) physical status II or III
* Scheduled for elective cesarean section
* Undergoing surgery under standardized spinal anesthesia

Exclusion Criteria:

* Pre-existing headache disorders (e.g., migraine, chronic tension-type headache)
* Known ophthalmic conditions (e.g., optic neuropathy, glaucoma)
* Inability to cooperate with ONSD(Optic Nerve Sheath Diameter) ultrasound measurements or follow-up
* Allergy to local anesthetics
* Emergency cesarean section
* Contraindications to spinal anesthesia:

  * Coagulopathy
  * Infection at the puncture site
* Preexisting hypertension on medication
* Pre-eclampsia with severe features (suggested for separate study)
* Known cardiac disease with hemodynamic instability
* Allergy to study drugs
* Fetal distress or non-reassuring cardiotocography (CTG)
* Body Mass Index (BMI) >40 kg/m²
* Refusal to sign informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Cesarean Section
Study Population: Target Population:
  The target population consists of adult female parturients who are medically eligible for spinal anesthesia and are undergoing elective cesarean delivery in a hospital setting.
  Source Population:
  The source population is defined as all consecutive adult female patients (aged 18-45 years, ASA II-III) who are admitted to Benha University Hospitals for an elective cesarean section during the study enrollment period (December 2025 - June 2026) and who meet the eligibility criteria.
  Study Sample (Final Cohort):
  The study sample will comprise 150 consenting patients drawn consecutively from the source population, forming a single observational cohort. These participants will undergo standardized spinal anesthesia and serial Optic Nerve Sheath Diameter (ONSD) measurements, with follow-up for Post-Dural Puncture Headache development over 72 hours.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Optimal Delta ONSD cut-off value for predicting PDPH | 72 hours post-spinal.
  To determine the numerical value of the change in Optic Nerve Sheath Diameter (Delta ONSD = ONSD<sub>pre</sub> - ONSD<sub>post</sub>) that best predicts the development of PDPH.

SECONDARY OUTCOMES:
Post-Dural Puncture Headache (PDPH) | 72h.
  To assess the intensity of headache pain. By Numeric Rating Scale (NRS):
  0 (no pain) to 10 (worst imaginable pain).
The Need for Epidural Blood Patch (EBP) | 72 hour
  The % of patients requiring an Epidural Blood Patch will de determined

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data could be shared upon a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP